CLINICAL TRIAL: NCT07265427
Title: Acceptance and Perceived Benefits of Digitalization by Medical Assistants and Other Generational Groups (ANDI-MFA-2): "Trust in AI and Digitalization in Healthcare Across Generational Groups: A Comparative Study of Barriers and Facilitators Toward Equitable Adoption"
Brief Title: Trust in AI and Digitalization in Healthcare Across Generational Groups: A Comparative Study of Barriers and Facilitators Toward Equitable Adoption.
Acronym: TRUST-AI
Status: Recruiting | Type: Observational
Sponsor: Jacobs University Bremen gGmbH (Other)
Collaborators: Hamburg University of Applied Sciences/Hochschule für Angewandte Wissenschaften Hamburg (HAW Hamburg) (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Sonia Lippke, Head of Health Psychology & Behavioral Medicine Unit, Jacobs University Bremen gGmbH
Other Study IDs: ANDI-MFA2
Record Dates: First submitted 2025-11-18; First posted 2025-12-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Digital Health; Artificial Intelligence (AI)
Keywords: Artificial Intelligence (AI); Digitalization; Trust; Barriers; Facilitators; Intergenerational Comparision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Rehabilitation Center Oldenburg patients and employees: Patients and employees at a rehabilitation center Oldenburg.
- training course participants: Seniors participating in "Digital in Old Age" training courses.
- Students: Students at HAW Hamburg

SUMMARY:
This study aims to investigate differences in perception of barriers and facilitators of digitalization and Artificial Intelligence (AI) usage in healthcare across different generational groups (youth, working-age adults, and seniors). The results will help create practical recommendations for public health projects and consultants to support fair and inclusive use of new digital tools in healthcare. A cross-sectional online survey will be conducted among students at HAW, patients and employees in the rehabilitation center in Oldenburg, and seniors participating in the "Digital im Alter"(DIA) project.

DETAILED DESCRIPTION:
This study will use an online questionnaire to collect data from respondents about their attitudes toward digital technologies and artificial intelligence in healthcare, as well as their opinions about barriers and facilitators for the equal adoption of modern technologies. The survey will be conducted in November to December 2025.

The survey will use validated scales, including the eHealth Literacy Scale (eHEALS) and the Human-Computer Trust Scale (HCTS), combined with additional items assessing perceived barriers and facilitators. Open-ended questions will allow participants to express their views on barriers and facilitators in their own words and from their perspective.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Belonging to one of the defined participant groups
* Consent to participate in the online survey
* Ability to participate in the survey (e.g., sufficient German or English language skills)

Exclusion Criteria:

* Individuals under 18
* Inability to give informed consent
* Illiteracy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population is chosen in a way that the cohorts can cover all three generations required for the comparative study. Therefore, the cohorts in this study are:
  * Students at Hamburg University of Applied Sciences.
  * Seniors participating in "Digital in Old Age" training courses.
  * Patients and employees at a rehabilitation center in Oldenburg.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Trust in digitalization and AI in healthcare | December 2025 - January 2026
  * Measured with the adapted Human-Computer Trust Scale (HCTS). Total scores are calculated by summing ten items rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree), resulting in a minimum possible score of 10 and a maximum of 50. Higher scores indicate a greater level of trust in the computer system or AI.
  * Comparison across generational groups (youth, working-age adults, seniors).
Perceived barriers to adoption of AI and digitalization in healthcare | December 2025 - January 2026
  * Measured with 5 Likert-scale items (accuracy, privacy and security, lack of human contact, ethics, lack of knowledge). Each item is rated from 1 = no concern to 5 = very strong concern.
  * Open-ended question: "What is your biggest concern about AI and digital technologies in healthcare and why?"
  * Comparison across generational groups (youths, working-age adults, seniors). Analysis of universal and generation-specific barriers.
Perceived facilitators to the adoption of AI and digitalization in healthcare | December 2025 - January 2026
  * Measured with 6 Likert-scale items (clear explanations, regulation, professional review, transparent data use, training, success stories). Each item is rated from 1 = not effective to 5 = very effective.
  * Open-ended question: "What would help you personally to trust in digital technologies and AI in healthcare?"
  * Comparison across generational groups (youths, working-age adults, seniors). Analysis of universal and generation-specific facilitators.

SECONDARY OUTCOMES:
eHealth literacy and digital skills | December 2025 - January 2026
  * Measured with the eHEALS (The eHealth Literacy Scale). Total scores are calculated by summing eight items rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree), resulting in a minimum possible score of 8 and a maximum of 40. Higher scores indicate better perceived eHealth literacy.
  * Descriptive analysis and role as a potential moderator of trust and acceptance across generational groups.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Constructor University (formerly known as Jacobs University), Bremen
  - HAW Hamburg, Hamburg

IPD SHARING:
Plan to Share IPD: No